CLINICAL TRIAL: NCT03235362
Title: A Phase 1, Randomized, Open-label, Multiple-dose, 3-treatment, 6-sequence, 3-period Crossover Clinical Trial to Investigate the Safety and Pharmacokinetic Drug Interaction Between YHR1705 and YHR1706 in Healthy Volunteers
Brief Title: A Clinical Trial to Investigate the Pharmacokinetic Drug Interaction Between YHR1705 and YHR1706
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YH14755-103
Record Dates: First submitted 2017-07-25; First posted 2017-08-01 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-07

CONDITIONS: Dyslipidemia; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1 (Experimental): 5 subjects will be assigned In this group. Subjects will receive multiple oral doses of YHR1705+YHR1706 QD for 5 consecutive days during period 1.
  Subjects will receive multiple oral doses of YHR1706 QD for 5 consecutive days during period 2.
  Subjects will receive multiple oral doses of YHR1705 QD for 5 consecutive days during period 3.
  Interventions: Drug: YHR1705; Drug: YHR1706; Drug: YHR1705+YHR1706
- 2 (Experimental): 5 subjects will be assigned In this group. Subjects will receive multiple oral doses of YHR1705 QD for 5 consecutive days during period 1.
  Subjects will receive multiple oral doses of YHR1705+YHR1706 QD for 5 consecutive days during period 2.
  Subjects will receive multiple oral doses of YHR1706 QD for 5 consecutive days during period 3.
  Interventions: Drug: YHR1705; Drug: YHR1706; Drug: YHR1705+YHR1706
- 3 (Experimental): 5 subjects will be assigned In this group. Subjects will receive multiple oral doses of YHR1706 QD for 6 consecutive days during period 1.
  Subjects will receive multiple oral doses of YHR1705 QD for 5 consecutive days during period 2.
  Subjects will receive multiple oral doses of YHR1705+YHR1706 QD for 5 consecutive days during period 3.
  Interventions: Drug: YHR1705; Drug: YHR1706; Drug: YHR1705+YHR1706
- 4 (Experimental): 5 subjects will be assigned In this group. Subjects will receive multiple oral doses of YHR1705 QD for 5 consecutive days during period 1.
  Subjects will receive multiple oral doses of YHR1706 QD for 6 consecutive days during period 2.
  Subjects will receive multiple oral doses of YHR1705+YHR1706 QD for 5 consecutive days during period 3.
  There will be a washout of at least 10 days between the last dose in one period and the first dose in the subsequent period.
  Interventions: Drug: YHR1705; Drug: YHR1706; Drug: YHR1705+YHR1706
- 5 (Experimental): 5 subjects will be assigned In this group. Subjects will receive multiple oral doses of YHR1706 QD for 5 consecutive days during period 1.
  Subjects will receive multiple oral doses of YHR1705+YHR1706 QD for 5 consecutive days during period 2.
  Subjects will receive multiple oral doses of YHR1705 QD for 5 consecutive days during period 3.
  Interventions: Drug: YHR1705; Drug: YHR1706; Drug: YHR1705+YHR1706
- 6 (Experimental): 5 subjects will be assigned In this group. Subjects will receive multiple oral doses of YHR1705+YHR1706 QD for 5 consecutive days during period 1.
  Subjects will receive multiple oral doses of YHR1705 QD for 5 consecutive days during period 2.
  Subjects will receive multiple oral doses of YHR1706 QD for 5 consecutive days during period 3.
  Interventions: Drug: YHR1705; Drug: YHR1706; Drug: YHR1705+YHR1706

INTERVENTIONS:
Drug: YHR1705 — Subjects will receive multiple oral doses of YHR1705 QD for 5 consecutive days in each period.
Drug: YHR1706 — Subjects will receive multiple oral doses of YHR1706 QD for 5 consecutive days in each period.
Drug: YHR1705+YHR1706 — Subjects will receive multiple oral doses of YHR1705 + YHR1706 QD for 5 consecutive days in each period.

SUMMARY:
This is a phase 1, open label, multiple-dose, crossover clinical trial to investigate the pharmacokinetic drug interaction between YHR1705 and YHR1706 in healty male volunteers

DETAILED DESCRIPTION:
This is an open-label, randomized, 6-sequence, 3-period crossover study. Subjects will receive multiple oral doses of YHR1705, YHR1706 or YHR1705 + YHR1706 QD for 5 consecutive days. There will be a washout of at least 10 days between the last dose in one period and the first dose in the subsequent period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male with body mass index(BMI) between 18.5 and 30 kg/m2
* Who has not suffered from clinically significant disease
* Provision of signed written informed consent

Exclusion Criteria:

* History of and clinically significant disease
* A history of drug abuse or the presence of positive reactions to drugs that have abuse potential in urine screenings for drugs
* Administration of other investigational products within 3 months prior to the first dosing
* Volunteers considered not eligible for the clinical trial by the investigator due to reasons including laboratory test results, ECGs, or vital signs

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male with body mass index (BMI) between 18.5kg/m2 and 30kg/m2
Enrollment: 28 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
YHR1705, YHR1706 AUCtau | 0 - 24hours
  AUCtau
YHR1705, YHR1706 Css, max | 0 - 24hours
  Css,max

CONTACTS AND LOCATIONS:
Overall Officials: Mingul Kim, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No